CLINICAL TRIAL: NCT03938558
Title: Art for MS - Effects of a 10 Week Multimodal Dance and Art Intervention Program on Fatigue, Fatigability, and Their Related Factors - A Controlled Pilot-trial
Brief Title: Art for MS - Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B9115201836892
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: multiple sclerosis; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Intervention Model Description: This study distinguish two groups contributing to a dance and art production. The experimental group will perform 10 weeks of dance training, while the other group will contribute to the production in various ways (e.g. word art, photography, painting, …).
  Measures will be taken before and after the training or assistance in the production.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance intervention group (Experimental): * Dancers at beginners level
  * Dancers at advanced level
  Interventions: Other: MS-Dance
- Art intervention group (Active Comparator): * Paint artists
  * Word artists
  * Film artists
  * Photographers
  Interventions: Other: MS-Art

INTERVENTIONS:
Other: MS-Dance — The experimental group will perform 10 weeks of dance training
  Arms: Dance intervention group
Other: MS-Art — The other group will contribute to the production in various ways (e.g. word art, photography, painting, …)
  Arms: Art intervention group

SUMMARY:
This study is a controlled pilot study with 17 participants with Multiple Sclerosis (MS). The primary goal of this study is to objectively examine the effects of a multimodal dance intervention on walking-related performance fatigability. The secondary aim is to investigate the effects of a multimodal dance intervention on other MS symptoms related to fatigue and fatigability.

The following research questions will be addressed:

1. Does a multimodal dance intervention have positive effects on walking-related fatigability?
2. Does a multimodal dance intervention have positive effects on other MS symptoms related to fatigue and fatigability?

DETAILED DESCRIPTION:
This study distinguish two groups contributing to a dance and art production. The experimental group will perform 10 weeks of dance training, while the other group will contribute to the production in various ways (e.g. word art, photography, painting, …).

Measures will be taken before and after the training or assistance in the production.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 70 years
* Confirmed diagnosis according to the McDonald criteria
* Able to walk independently or with bilateral support for 6 minutes
* Signed the informed consent

Exclusion Criteria:

* Exacerbation or relapse within last 3 months before onset study
* Other medical conditions interfering with walking ability (e.g. cardiac or respiratory diseases, arthritis, fibromyalgia, Parkinson and stroke)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
motor fatigability | Baseline
  Performance motor fatigability: Calculating the Distance Walked Index (DWI) during 6MWT.
  Formula for walking-related performance fatigability: DWI = ([Distance walked at minute 6 - Distance walked at minute 1]/Distance walked at minute 1) × 100
motor fatigability | week 10
  Performance motor fatigability: Calculating the Distance Walked Index (DWI) during 6MWT.
  Formula for walking-related performance fatigability: DWI = ([Distance walked at minute 6 - Distance walked at minute 1]/Distance walked at minute 1) × 100
motor fatigability | week 20
  Performance motor fatigability: Calculating the Distance Walked Index (DWI) during 6MWT.
  Formula for walking-related performance fatigability: DWI = ([Distance walked at minute 6 - Distance walked at minute 1]/Distance walked at minute 1) × 100
Trait motor fatigue | baseline
  Modified Fatigue Impact Scale (MFIS)
Trait motor fatigue | week 10
  Modified Fatigue Impact Scale (MFIS)
Trait motor fatigue | week 20
  Modified Fatigue Impact Scale (MFIS)

SECONDARY OUTCOMES:
Coördination test with lower limbs | baseline
  seated bipedal coordination task (knee flexion and extension movements during 6 minutes, and metronome based 0,75 Hz, 1Hz and 1,5 Hz for 1 minute)
Coördination test with lower limbs | week 10
  seated bipedal coordination task (knee flexion and extension movements during 6 minutes, and metronome based 0,75 Hz, 1Hz and 1,5 Hz for 1 minute)
Coördination test with lower limbs | week 20
  seated bipedal coordination task (knee flexion and extension movements during 6 minutes, and metronome based 0,75 Hz, 1Hz and 1,5 Hz for 1 minute)
Perceived motor fatigability | Baseline
  VAS increase minute per minute during 6MWT (range 0-10)
Perceived motor fatigability | week 10
  VAS increase minute per minute during 6MWT (range 0-10)
Perceived motor fatigability | week 20
  VAS increase minute per minute during 6MWT (range 0-10)
Performance cognitive fatigability and cognitive capacity | Baseline
  PASAT and SDMT total score and correct answers last ⅓ vs first ⅓
Performance cognitive fatigability and cognitive capacity | week 10
  PASAT and SDMT total score and correct answers last ⅓ vs first ⅓
Performance cognitive fatigability and cognitive capacity | week 20
  PASAT and SDMT total score and correct answers last ⅓ vs first ⅓
Trait fatigue | Baseline
  Fatigue Severity Scale (FSS) : range 1-7
Trait fatigue | week 10
  Fatigue Severity Scale (FSS) : range 1-7
Trait fatigue | week 20
  Fatigue Severity Scale (FSS) : range 1-7
MSIS-29 Questionnaire | Baseline
  Impact of MS via a questionnaire. 29 items, total score on 145.
MSIS-29 Questionnaire | week 10
  Impact of MS via a questionnaire. 29 items, total score on 145.
MSIS-29 Questionnaire | week 20
  Impact of MS via a questionnaire. 29 items, total score on 145.
SF-36 Questionnaire | Baseline
  Quality of Life health related questionnaire. Scale 0-100
SF-36 Questionnaire | week 10
  Quality of Life health related questionnaire. Scale 0-100
SF-36 Questionnaire | week 20
  Quality of Life health related questionnaire. Scale 0-100
ABC scale | Baseline
  Activity balance confidence scale. Scale has 16 items and is transferred to a percentage.
ABC scale | week 10
  Activity balance confidence scale. Scale has 16 items and is transferred to a percentage.
ABC scale | week 20
  Activity balance confidence scale. Scale has 16 items and is transferred to a percentage.
MSWS-12 Questionnaire | Baseline
  Questionnaire about walking in MS, 12 items, total score on 60, minimum score 12.
MSWS-12 Questionnaire | week 10
  Questionnaire about walking in MS, 12 items, total score on 60, minimum score 12.
MSWS-12 Questionnaire | week 20
  Questionnaire about walking in MS, 12 items, total score on 60, minimum score 12.
5xSTS T25FW | Baseline
  5 times sit to stand test, where patients have to stand and sit 5 times as fast as possible. Determined in seconds
5xSTS T25FW | week 10
  5 times sit to stand test, where patients have to stand and sit 5 times as fast as possible. Determined in seconds
5xSTS T25FW | week 20
  5 times sit to stand test, where patients have to stand and sit 5 times as fast as possible. Determined in seconds
T25FW test | Baseline
  patients have to walk 25 feet as fast as possible. Determined in seconds
T25FW test | week 10
  patients have to walk 25 feet as fast as possible. Determined in seconds
T25FW test | week 20
  patients have to walk 25 feet as fast as possible. Determined in seconds
NHPT (Nine hole peck test) | Baseline
  Nine hole peck test: descriptive measure for hand dexterity. Measured in seconds.
NHPT (Nine hole peck test) | week 10
  Nine hole peck test: descriptive measure for hand dexterity. Measured in seconds.
NHPT (Nine hole peck test) | week 20
  Nine hole peck test: descriptive measure for hand dexterity. Measured in seconds.
DGI (Dynamic gait index) | Baseline
  patient have to perform several static and dynamic balance test. A four-point ordinal scale, ranging from 0-3. "0" indicates the lowest level of function and "3" the highest level of function. Total Score = 24
DGI (Dynamic gait index) | week 10
  patient have to perform several static and dynamic balance test. A four-point ordinal scale, ranging from 0-3. "0" indicates the lowest level of function and "3" the highest level of function. Total Score = 24
DGI (Dynamic gait index) | week 20
  patient have to perform several static and dynamic balance test. A four-point ordinal scale, ranging from 0-3. "0" indicates the lowest level of function and "3" the highest level of function. Total Score = 24
EmNSA | Baseline
  Dynamic gait index: patient have to perform several static and dynamic balance test. A ordinal scale, ranging from 0-2. "0" indicates the lowest level of function and "2" the highest level of function. Total Score = 48
EmNSA | week 10
  Dynamic gait index: patient have to perform several static and dynamic balance test. A ordinal scale, ranging from 0-2. "0" indicates the lowest level of function and "2" the highest level of function. Total Score = 48
EmNSA | week 20
  Dynamic gait index: patient have to perform several static and dynamic balance test. A ordinal scale, ranging from 0-2. "0" indicates the lowest level of function and "2" the highest level of function. Total Score = 48
CMI (Cognitive motor interference) | Baseline
  Dual task testing during 1 min tasks and 6 minutes task to measure alertness of movement control.
  Dual task testing during 1 min tasks and 6 minutes task to measure alertness of movement control.
CMI (Cognitive motor interference) | week 10
  Dual task testing during 1 min tasks and 6 minutes task to measure alertness of movement control.
  Dual task testing during 1 min tasks and 6 minutes task to measure alertness of movement control.
CMI (Cognitive motor interference) | week 20
  Dual task testing during 1 min tasks and 6 minutes task to measure alertness of movement control.
  Dual task testing during 1 min tasks and 6 minutes task to measure alertness of movement control.

CONTACTS AND LOCATIONS:
Overall Officials: peter Feys, prof. dr., Principal Investigator — Hasselt University; Fanny Van Geel, drs., Study Chair — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium

REFERENCES:
- [Derived] Goetschalckx M, Van Geel F, Meesen R, Triccas LT, Geraerts M, Moumdjian L, Feys P. Interlimb Coordination Performance in Seated Position in Persons With Multiple Sclerosis: Reduced Amplitude Over 6 min and Higher Coordination Variability in Persons With Walking Fatigability. Front Hum Neurosci. 2021 Oct 20;15:765254. doi: 10.3389/fnhum.2021.765254. eCollection 2021. PMID 34744669